CLINICAL TRIAL: NCT01559012
Title: The CLONEMESI Study: a Randomized Placebo-controlled Study With Transdermal Clonidine in the Treatment of Severe Hyperemesis Gravidarum.
Brief Title: Transdermal Clonidine in the Treatment of Severe Hyperemesis Gravidarum
Acronym: CLONEMESI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Aldo Maina, M.D. Unit of Obstetric Medicine. Principal Investigator, Azienda Ospedaliera Ospedale Infantile Regina Margherita Sant'Anna
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Registro CE 409 det. 163/2012
Record Dates: First submitted 2012-03-12; First posted 2012-03-20 (Estimated); Results first posted 2014-04-30 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-03

CONDITIONS: Hyperemesis Gravidarum
Keywords: Hyperemesis Gravidarum; treatment; transdermal clonidine
MeSH Terms: conditions — Hyperemesis Gravidarum | interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- clonidine first - placebo second (Other): in this group patients are treated with transdermal clonidine first for 5 days then switch to placebo for 5 days
  Interventions: Drug: Clonidine
- placebo first - clonidine second (Other): in this group patients are treated with placebo first for 5 days then with transdermal clonidine for next 5 days
  Interventions: Drug: Clonidine

INTERVENTIONS:
Drug: Clonidine — transdermal clonidine patch 5 mg q. 5 days
  Other Names: Catapresan TTS 2 transdermal patch

SUMMARY:
CLONEMESI is an academic, independent, randomized placebo-controlled trial to assess the effect of transdermal (TD) clonidine in improving the symptoms of severe Hyperemesis Gravidarum(HG) affecting women in their 6th-12th week of pregnancy. The study has a crossover design.

DETAILED DESCRIPTION:
Setting. The trial is performed at a single hospital setting after admission of patients.

Ethics. The study has been approved by our local Ethics Committee and women are requested to sign an informed consent. No pharmaceutical company is involved in any phases of the trial including protocol design, study conduction, coordination and monitoring, data handling and analysis.

Randomization. The patients are allocated to a random list to receive first placebo and then TD clonidine or the other way round.

Blinding. Neither the patients nor their attending caregivers know the order of administration . The outcome assessors are blinded as well.

Treatment.The patients are randomly treated with and without TD clonidine for 2 consecutive periods of 5 days , other antiemetic drugs (promethazine, metoclopramide, ondansetron) and anti- reflux drugs (ranitidine, omeprazole) being administered on a scheduled or as-needed basis. All patients receive intravenous hydration and supplementation with thiamine.

Assessment. Physical condition of patients are assessed daily: blood pressure (lying and standing), body weight, morning ketonuria. Two different clinical self administered scores as PUQE (Pregnancy Unique Quantification of Emesis) and VAS (Visual Analogue Scale) are employed to check daily the intensity of symptoms and the sense of wellbeing. The consumption of antiemetic and anti-reflux drugs administered in the two periods is monitored .

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 6-12 weeks and a major grade of HG clinical severity defined as follows:
* a PUQE score index ≥ 13 associated to one or more of the following conditions:
* weight loss > 5% of pregravidic weight,
* electrolyte disturbances,
* dehydration,
* duration of symptoms > 10 days ,
* inadequate food and drink intake

Exclusion Criteria:

* Language barrier.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Maina, M.D., Principal Investigator — Dipartimento di Ostetricia e Neonatologia. Servizio di Medicina Interna. Ospedale Sant'Anna Torino; Tullia Todros, M.D., Study Chair — Head . Dipartimento di Ostetricia e Neonatologia. Università di Torino.
Locations (1):
- Ospedale Sant'Anna. Dipartimento di Ostetricia e Neonatologia. Servizio di Medicina Interna, Torino, Italy

REFERENCES:
- [Derived] Maina A, Arrotta M, Cicogna L, Donvito V, Mischinelli M, Todros T, Rivolo S. Transdermal clonidine in the treatment of severe hyperemesis. A pilot randomised control trial: CLONEMESI. BJOG. 2014 Nov;121(12):1556-62. doi: 10.1111/1471-0528.12757. Epub 2014 Apr 1. PMID 24684734

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients admitted to hospital for severe hyperemesis (HG) March - December 2012
Pre-assignment Details: The crossover study design allows to compare in the same patient the response to different treatment schedules.
  The assumption is that the condition treated is not changing over the time of observation.
  The reported evidence in literature is that severe HG does not spontaneously improve till 14th week.
Groups:
- Clonidine First - Placebo Second: in this group patients are treated with TD clonidine first for 5 days then switch to placebo for 5 days
  Clonidine : transdermal clonidine patch 5 mg q. 5 days
- Placebo First - Clonidine Second: in this group patients are treated with placebo first for 5 days then with TD clonidine for next 5 days
  Clonidine : transdermal clonidine patch 5 mg q. 5 days
Period: Overall Study
Arm/Group | Clonidine First - Placebo Second | Placebo First - Clonidine Second
Started | 6 | 7 (1 more patient added to randomization list to reach the pre-assignment number of treated patients)
Completed | 6 | 6 (Patient N. 2 withdrew from study for alleged side effects at day 1 of placebo cycle.)
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline biophysical and demographic data were reported:
  age, race, ethnicity, parity, HG in previous pregnancy, smoking, BMI, weight loss, concurrent diseases, concurrent treatment,gestational age at start of symptoms, gestational age at enrollment, PUQE score at enrollment
Groups:
- Total: Total of all reporting groups
Arm/Group | Clonidine First - Placebo Second | Placebo First - Clonidine Second | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 13
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (5.46) | 32.3 (5.99) | 32.1 (5.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: PUQE Score for Assessment of Severity in Hyperemesis Gravidarum
Description: PUQE in an acronym for Pregnancy Unique Quantification of Emesis, a validated clinical score for assessment of severity of emesis in pregnancy.
  It is composed of three items; every item has a score from 1 (best) to 5 (worst).
  The sum range varies from 3 (best) to 15 (worst). Participants are followed for the whole duration of hospital stay (10 days) asking them to score their symptoms daily.
Time Frame: Mean values of first period of five days are compared with mean values of second period of five days. Change is reported as baseline value - value at day 5 or at day 10.
Population: A sample size calculation for crossover studies using a model available on line (MGH Mallinckrodt General Clinical Research Center - Harvard Medical School) showed that a total of 12 patients were needed in order to detect a difference of 2 points of PUQE score between the two groups at P < 0.01 and a beta > 0.90.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Clonidine: Six patients are treated with TD clonidine first for 5 days then switch to placebo for next 5 days Other six patients are treated with placebo first, for 5 days, then are switched to TD clonidine for next 5 days.
  The allocation order for every patient is randomized.
  Every patient is the comparison as to herself
- Placebo: Six patients are treated with TD clonidine first,for 5 days, then switch to placebo for next 5 days Other six patients are treated with placebo first, for 5 days, then are switched to TD clonidine for next 5 days.
  The allocation order for every patient is randomized
  Every patient is the comparison as to herself
Arm/Group | Clonidine | Placebo
Number analyzed (Participants) | 12 | 12
units on a scale | 6.3 (5.5-7.11) [5.5 to 7.1] | 8.5 (7.3-9.3) [7.7 to 9.3]
Statistical Analysis 1: Comparison: Clonidine vs Placebo; This is an analysis between groups of intervention clonidine versus placebo. Statistical signiﬁcance was assessed by the use of Mann-Whitney U test P < 0.05 was deﬁned as statistically signiﬁcant . Data are presented as mean + SD; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney) — A sample size modeling (MGH Mallinckrodt General Clinical Research Center) showed that a total of 12 patients were needed in order to detect a difference of 2 points of PUQE score between the two groups at P < 0.01 and a beta > 0.90; Statistical signiﬁcance was assessed by the use of Mann-Whitney U test. P < 0.05 was deﬁned as statistically signiﬁcant; Mean Difference (Final Values) = 2.2, 95% CI 2-sided [1.05 to 3.32], Standard Deviation 2.7
Statistical Analysis 2: Comparison: Clonidine vs Placebo; This is a within patient variation between clonidine and placebo. Statistical signiﬁcance was assessed by the use of Mann-Whitney U test P < 0.05 was deﬁned as statistically signiﬁcant . Data are presented as mean +/- Standard Deviation (SD); Test type: Non-Inferiority or Equivalence — A sample size modeling (MGH Mallinckrodt General Clinical Research Center) showed that a total of 12 patients were needed in order to detect a difference of 2 points of PUQE score between the two groups at P < 0.01; p < 0.02, Wilcoxon (Mann-Whitney); within patient variation = 1.83, 95% CI 2-sided [0.43 to 3.24]

2. Primary Outcome: VAS Score for Assessment of Severity in Hyperemesis Gravidarum
Description: VAS is a Visual Analogic Scale formulated in 5 items. Every item has a score from 0 (best) to 10 (worst). The sum range swings from 0 (best ) to 50 (worst). Participants are followed for the whole duration of hospital stay (10 days) asking them to score their symptoms daily.
Time Frame: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Clonidine: in this group patients are treated with TD clonidine first for 5 days then switch to placebo for 5 days
  Clonidine : transdermal clonidine patch 5 mg q. 5 days
- Placebo: in this group patients are treated with placebo first for 5 days then with TD clonidine for next 5 days
  Clonidine : transdermal clonidine patch 5 mg q. 5 days
Arm/Group | Clonidine | Placebo
Number analyzed (Participants) | 12 | 12
units on a scale | 22 [19 to 26] | 29 (2.58) [25 to 32]
Statistical Analysis 1: Comparison: Clonidine vs Placebo; Analysis within groups clonidine versus placebo. Statistical signiﬁcance was assessed by the use of Mann-Whitney U test P < 0.05 was deﬁned as statistically signiﬁcant . Data are presented as mean + SD; Test type: Superiority or Other; p = 0.009, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 7, 95% CI 2-sided [1.78 to 11.5]
Statistical Analysis 2: Comparison: Clonidine vs Placebo; Analysis within-patient. Statistical signiﬁcance was assessed by the use of Mann-Whitney U test P < 0.05 was deﬁned as statistically signiﬁcant . Data are presented as mean + SD; Test type: Non-Inferiority or Equivalence — A sample size modeling for crossover studies (MGH Mallinckrodt General Clinical Research Center) showed that a total of 12 patients were needed in order to detect a difference of 2 points of PUQE score between the two groups at P < 0.01; p < 0.01, Wilcoxon (Mann-Whitney); within patient variation = 7.5, 95% CI 2-sided [2.17 to 12.83]

3. Secondary Outcome: Morning Urine Ketonuria
Description: Morning urine ketonuria is a simple direct marker of starving associated to nausea and vomiting
Time Frame: participants are followed for the whole duration of hospital stay (10 days) comparing the first period of 5 days with the second period of 5 days
Measure: Mean (95% Confidence Interval); unit: Proportion of person-days
Groups:
- Clonidine; Placebo: All patients were treated with TD clonidine for 5 days and switched to placebo for 5 days, or the other way round
  Allocation order randomized
Arm/Group | Clonidine | Placebo
Number analyzed (Participants) | 12 | 12
Proportion of person-days | 0.06 [0.04 to 0.18] | 0.36 [0.24 to 0.47]
Statistical Analysis 1: Comparison: Clonidine vs Placebo; All patients were treated with TD clonidine for 5 days and switched to placebo for 5 days, or the other way round Allocation order randomized; Test type: Superiority or Other; p = 0.000, Wilcoxon (Mann-Whitney); difference of percentage of positivity = 0.30, 95% CI 2-sided [0.04 to 0.47]

4. Secondary Outcome: Daily Doses of Standard Antiemetic Drugs Required in the Two Different Periods.
Description: The patients were randomly treated with and without TD clonidine (5mg patch) for 2 consecutive periods of 5 days , other antiemetic drugs (promethazine, prochlorperazine, metoclopramide, ondansetron) and anti reflux drugs (ranitidine, omeprazole) being administered on a scheduled or as-needed basis.
  All patients received intravenous hydration and supplementation with thiamine, during both periods. The use of steroids was allowed as a rescue medication in case of further worsening of symptoms.
Time Frame: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: daily doses of antiemetics
Groups:
- Clonidine: All patients were treated with TD clonidine for 5 days and switched to placebo for 5 days, or the other way round
- Placebo: All patients were treated with TD clonidine for 5 days and switched to placebo for 5 days, or the other way round
  Clonidine : transdermal clonidine patch 5 mg q. 5 days
Arm/Group | Clonidine | Placebo
Number analyzed (Participants) | 12 | 12
daily doses of antiemetics | 1.5 [1.1 to 2.9] | 2.3 [1.9 to 3.0]
Statistical Analysis 1: Comparison: Clonidine vs Placebo; Statistical signiﬁcance was assessed by the use of Mann-Whitney U test P < 0.05 was deﬁned as statistically signiﬁcant . Data are presented as mean + SD; Test type: Superiority or Other; p = 0.013, Wilcoxon (Mann-Whitney); mean values = 0.8, 95% CI 2-sided [0.13 to 1.57]

5. Secondary Outcome: Number of Days Off i.v. Therapy, the TD System (Clonidine/Placebo) Being Applied Only
Description: if the symptoms improve the patient and her doctors may decide to stop parenteral drugs continuing the TD system therapy.
Time Frame: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Proportion of person-days
Groups:
- Placebo: All patients were treated with TD clonidine for 5 days and switched to placebo for 5 days, or the other way round
Arm/Group | Clonidine | Placebo
Number analyzed (Participants) | 12 | 12
Proportion of person-days | 0.40 [0.28 to 0.54] | 0.20 [0.09 to 0.36]
Statistical Analysis 1: Comparison: Clonidine vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.051, Wilcoxon (Mann-Whitney); days off-therapy % = 29

6. Secondary Outcome: Number of Patients Choosing Active Treatment for Off-label, Compassionate Use.
Description: the patients were asked to choose between two transdermal systems (active drug versus placebo) as the most effective
Time Frame: at 10 days since start of treatment
Population: no determination of sample size
Measure: Number; unit: participants
Arm/Group | Clonidine | Placebo
Number analyzed (Participants) | 12 | 12
participants | 9 | 3
Statistical Analysis 1: Comparison: Clonidine vs Placebo; Test type: Superiority or Other; p = 0.0089, Fisher Exact; proportion = 0

7. Secondary Outcome: Pregnancy Outcome Measures: Birth Weight.
Description: Birth weight adjusted for gestational age at delivery is a measure of pregnancy outcome after treatment of HG.
Time Frame: at delivery
Population: no determination of sample size Recording for safety issue
Measure: Mean (Full Range); unit: grams
Groups:
- Mean Birth Weight of 12 Patients: All patients were treated with TD clonidine for 5 days and switched to placebo for 5 days, or the other way round
  Allocation order randomized
Arm/Group | Mean Birth Weight of 12 Patients
Number analyzed (Participants) | 12
grams | 3312 [2510 to 4180]

8. Secondary Outcome: Newborn Outcome Measure: APGAR Score.
Description: The APGAR score is the most common indicator of neonatal status immediately after delivery.
  The test is done by a doctor, midwife, or nurse. The health care provider will examine the baby's:
  Breathing effort Heart rate Muscle tone Reflexes Skin color Each category is scored with 0, 1, or 2, depending on the observed condition. The APGAR rating is based on a total score of 1 to 10. The higher the score, the better the baby is doing after birth.
Time Frame: at 1 minute and at 5 minutes after delivery
Population: APGAR score of newborns at 1 minute and at 5 minutes
Measure: Mean (Full Range); unit: units on a scale
Groups:
- APGAR Score at 1'; APGAR Score at 5': All patients were treated with TD clonidine for 5 days and switched to placebo for 5 days, or the other way round
Arm/Group | APGAR Score at 1' | APGAR Score at 5'
Number analyzed (Participants) | 12 | 12
units on a scale | 9 [9 to 9] | 9 [9 to 9]

9. Secondary Outcome: Systolic Blood Pressure
Description: Systolic BP was measured every day during the clonidine treatment (5 days) and placebo (5 days)
Time Frame: 10 days
Measure: Mean (95% Confidence Interval); unit: mmHg
Groups:
- Clonidine: systolic blood pressure was recorded during clonidine treatment cycle
- Placebo: systolic blood pressure was recorded during placebo cycle
Arm/Group | Clonidine | Placebo
Number analyzed (Participants) | 12 | 12
mmHg | 91 [87 to 94] | 97 [93 to 100]
Statistical Analysis 1: Comparison: Clonidine vs Placebo; Test type: Superiority or Other; p = 0.01, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 6, 95% CI 2-sided [0.9 to 10.9]

10. Secondary Outcome: Diastolic Blood Pressure
Description: Diastolic BP was recorded every day during clonidine (5 days) and placebo (5 days) cycle
Time Frame: 10 days
Measure: Mean (95% Confidence Interval); unit: mmHg
Groups:
- Clonidine: diastolic blood pressure was recorded every day during clonidine treatment cycle
- Placebo: diastolic blood pressure was recorded every day during placebo cycle
Arm/Group | Clonidine | Placebo
Number analyzed (Participants) | 12 | 12
mmHg | 58 [55 to 60] | 61 [59 to 63]
Statistical Analysis 1: Comparison: Clonidine vs Placebo; Test type: Superiority or Other; p = 0.055, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 3, 95% CI 2-sided [0.3 to 6.3]

ADVERSE EVENTS:
Time Frame: 10 days of hospital stay
Description: For 5 days the patient received TD clonidine, the other 5 days received placebo.
Groups:
- Clonidine: patients are treated with transdermal clonidine patch 5 mg for 5 days
- Placebo: patients are treated with placebo (sham patch) for 5 days
Arm/Group | Clonidine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 0/6 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clonidine (N=6) | Placebo (N=7)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Itching was reported at day 1 on site of application of sham patch

LIMITATIONS AND CAVEATS:
Efficacy and safety issues are represented by maternal exposure in a critical period for organogenesis and hypotensive effect of the drug.

Findings based on a very limited number of women limit the reliability of results

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No